CLINICAL TRIAL: NCT06721429
Title: The Effect of Dual-task Training on Balance, Exercise Capacity, Cognitive Status, and Quality of Life in Individuals With Type 2 Diabetes Mellitus
Brief Title: The Effect of Dual-task Training on Balance, Exercise Capacity, Cognitive Status, and Quality of Life
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bartın Unıversity (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Gizem Mermerkaya, lecturer, Bartın Unıversity
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BARU-FTR-GM-02
Record Dates: First submitted 2024-12-03; First posted 2024-12-06 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: exercise; balance; exercise tolerance; Mental Status
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Motor Activity

STUDY DESIGN:
Intervention Model Description: This study will include 36 patients with type 2 diabetes mellitus. Patients who meet the inclusion criteria will be randomly assigned to one of three groups: the dual-task exercise training group (n=12), the single-task exercise training group (n=12), or the control group (n=12).In the single-task exercise training group, aerobic exercise, resistance training, and balance training will be performed as separate tasks, while in the dual-task training group, these same exercises will be performed simultaneously with cognitive dual-task training. The control group will be instructed to continue with their daily activities and refrain from participating in any exercise training program for eight weeks after the initial assessment. In the exercise training groups, individuals will undergo a combined exercise program consisting of aerobic exercise, resistance training, and balance training, with three sessions per week on non-consecutive days over a period of 8 weeks, totaling 24 sessions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- dual task exercise group (Experimental): Patients in the dual-task training group will undergo 60-minute conventional physiotherapy sessions three times a week for 8 weeks. Each physiotherapy session will consist of aerobic exercise, strengthening exercises, and balance training. In addition, cognitive exercise training will be incorporated into each session, performed concurrently with the conventional physiotherapy. The cognitive exercises provided in this study are structured to target areas such as memory, verbal fluency, executive functions, calculation, and attention.
  Interventions: Other: dual task exercise group
- single task exercise group (Active Comparator): Patients in the single-task training group will undergo 60-minute conventional physiotherapy sessions three times a week for 8 weeks. Each physiotherapy session will consist of aerobic exercise, strengthening exercises, and balance training.
  Interventions: Other: single task group
- control group (No Intervention): The control group will be instructed to continue with their daily activities and refrain from participating in any exercise training program for eight weeks after the initial assessment. After the exercise training period, the control group will also be invited to join the exercise training program of their choice.

INTERVENTIONS:
Other: dual task exercise group — Dual task exercise group Patients in the dual-task training group will undergo 60-minute conventional physiotherapy sessions three times a week for 8 weeks. Each physiotherapy session will consist of aerobic exercise, strengthening exercises, and balance training. In addition, cognitive exercise training will be incorporated into each session, performed concurrently with the conventional physiotherapy. The cognitive exercises provided in this study are structured to target areas such as memory, verbal fluency, executive functions, calculation, and attentioN Single task exercise group Patients in the single-task training group will undergo 60-minute conventional physiotherapy sessions three times a week for 8 weeks. Each physiotherapy session will consist of aerobic exercise, strengthening exercises, and balance training.
  Arms: dual task exercise group
Other: single task group — Single task exercise group Patients in the single-task training group will undergo 60-minute conventional physiotherapy sessions three times a week for 8 weeks. Each physiotherapy session will consist of aerobic exercise, strengthening exercises, and balance training.
  Arms: single task exercise group

SUMMARY:
The aim of this study is to investigate the effects of dual-task training on balance, exercise capacity, cognitive function, and quality of life in individuals with Type 2 Diabetes Mellitus (DM). As a result of this study, it is hoped that dual-task training will be an alternative to single-task training in the rehabilitation of individuals with Type 2 DM, with the goal of preventing falls and supporting a more active lifestyle. Additionally, it is intended to include dual-task training in preventive physiotherapy approaches. The main questions the study aims to answer are as follows:

Is dual-task training, conducted concurrently with exercise training, more effective in improving balance when compared to exercise training alone and the control group?

Is dual-task training, conducted concurrently with exercise training, more effective in improving exercise capacity, cognitive function, and quality of life when compared to exercise training alone and the control group?

The researchers will compare the effects of dual-task training in individuals with Type 2 diabetes by comparing the participants in the single-task exercise training group and the control group. Participants will be randomized into the dual-task exercise training group, the single-task exercise training group, and the control group. Individuals in the training group will undergo exercise training three days a week for 8 weeks.

DETAILED DESCRIPTION:
Geriatric individuals with Type 2 DM experience balance, gait, and cognitive impairments. Type 2 DM has been found to be associated with a 1.5 to 2.5-fold increased risk of dementia in the elderly population. In individuals with Type 2 DM, cognitive decline risk is heightened due to factors such as insulin resistance, impaired glucose metabolism, advanced glycation end-products, impaired amyloid beta degradation, increased oxidative stress, and inflammation. Among adults with Type 2 DM, the global prevalence of cognitive impairment is approximately 45%, with rates varying between 21.8% and 67.5% in different countries. Type 2 DM is most commonly linked to declines in episodic memory, verbal fluency, working memory, processing speed, and executive functions. Executive functions are "higher-level" processes that oversee and control other cognitive functions. These capabilities underpin activities such as planning, decision-making, switching between tasks, goal-directed behavior, and coordinating ongoing activities (e.g., multitasking or planning a series of activities). More importantly, executive function is critical for sensory integration used to coordinate balance and gait motor output. Declines in executive function serve as a risk factor for falls in geriatric individuals with DM. Dual-task paradigms are used to examine the degree of automaticity of movement. In these paradigms, a primary task, often walking, is undertaken with the main focus on attention. Secondary tasks are added, and the effects on both tasks are evaluated. In everyday situations, such as walking and talking, it is common to perform multiple tasks simultaneously, thus these situations are essentially dual-task paradigms. When the combined load of two or more tasks exceeds available attention capacity, performance on one or both tasks will deteriorate. Impairments in executive function lead to the emergence of dual-task paradigms. These tasks can be motor-cognitive, cognitive-cognitive, or motor-motor. A previous study observed a negative impact of dual-tasking on gait parameters in individuals with Type 2 DM. This suggests that impaired dual-task capacity in Type 2 DM may contribute to the higher incidence of falls in this population. This highlights the need for training that develops the relationship between cognitive abilities and motor skills when planning rehabilitation programs. In studies conducted on other high-fall-risk groups (stroke survivors, Parkinson's disease, and elderly individuals with a fall history), the effects of dual-task training on balance have been described. Improvements in balance were explained by physical parameters such as gait speed and step length. However, since cognitive factors significantly influence balance, in addition to physical components, it is necessary to investigate the underlying cognitive functions of balance following dual-task training. In a study of elderly adults with a history of falls, it was shown that dual-task training was effective in improving both balance and executive function. It is believed that improvements in executive function in elderly individuals may be an effective way to enhance balance. A 2023 meta-analysis showed that combined exercise training (aerobic + resistance) improved cognitive function, particularly executive function, in individuals with Type 2 DM. Studies conducted on healthy adults have demonstrated that participation in simultaneous combined exercise and cognitive training (dual-task training) improves cognition beyond the effects of the individual components. These combined effects may have an additional impact on brain and physiological functions. While many studies in the literature have shown the positive effects of combined exercise on executive function in Type 2 DM, there are few studies investigating whether dual-task training, which has shown positive effects in other populations, is more effective in improving balance and executive function in individuals with Type 2 DM. A 2018 study demonstrated that step training exercises were feasible and improved executive function in adults with Type 2 DM and cognitive complaints. However, the effect of dual-task training combined with aerobic, strength, and balance exercises in individuals with Type 2 DM has not been previously investigated.

The aim of this study is to investigate the effects of dual-task training on balance, exercise capacity, cognitive function, and quality of life in individuals with Type 2 DM. This project will focus on dual-task training in geriatric individuals with Type 2 DM. The effects of cognitive exercises combined with exercise training will be compared with combined exercise training alone, focusing on balance, aerobic capacity, cognitive function, and quality of life. One of the complications in geriatric individuals with Type 2 DM is the decline in dual-task performance, which leads to deviations in normal gait, difficulties in maintaining balance, and ultimately mobility restrictions. It is expected that dual-task training will enhance dual-task performance more than single-task training. Investigators anticipate that this improvement in performance will allow geriatric individuals to spend more independent time in daily activities, enhance their balance, and improve their quality of life. Unlike conventional physiotherapy approaches, dual-task training aims to improve both motor and cognitive performance simultaneously, thus saving time. It is expected that participation in different and engaging exercise training will increase exercise participation (sustainability) in the short and/or long term. Investigators expect that dual-task training in geriatric individuals with Type 2 DM will improve cognitive performance, contribute to functional capacity, and prevent falls.

ELIGIBILITY:
Inclusion Criteria:

* Being followed up with a diagnosis of Type 2 Diabetes Mellitus for at least 6 months (fasting plasma glucose of 7.0 mmol/L or higher)
* Not having participated in any structured exercise program for at least 6 months prior.
* Being willing to volunteer for the study

Exclusion Criteria:

* Nephropathy
* Retinopathy
* Having dementia or Alzheimer's disease
* Using a walking aid
* Having ulceration
* Using balance-curing drugs
* Surviving myocardial infarction at least 6 months ago
* Stable or unstable angina pectoris
* Left ventricular ejection fraction below 40%
* Peripheral arterial diseases
* Resting blood pressure above 160/100 mmHg
* Body mass index above 35 kg/m2
* Having a history of deep vein thrombosis, pulmonary embolism or stroke in the past

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-12-25 (Estimated); Primary Completion 2025-02-03 (Estimated); Study Completion 2025-05-28 (Estimated)

PRIMARY OUTCOMES:
Time Up and Go Test | In 2 weeks
  This test is applied to assess the risk of falling and mobility.This test starts with the individual leaving the chair without receiving arm support by giving the go command while sitting in a chair.The distance of 3 meters is asked to return and sit again in the chair.The elapsed time is recorded in seconds.
Berg Balance Scale | In 2 weeks
  It is a 14-item scale that evaluates the tasks used in daily life activities.Standing up without support, standing without support, sitting without support, standing up, transfers, standing with feet, standing with legs while standing, reaching out while standing, picking up from the ground, looking back, 360 degree rotation, firm side standing on the stool, one foot standstill and standstill functions are evaluated.

SECONDARY OUTCOMES:
Functional Reaching Test | In 2 weeks
  The individual's limits of stability will be assessed by measuring the distance of forward reach while standing still. Prior to the assessment, a 122 cm tape measure will be attached to the wall at the level of the participant's acromion. The participant will be instructed to raise their right arm to 90° of flexion and make a fist. Initially, the starting point, marked by the position of the participant's 3rd metacarpal, will be measured and recorded. The participant will then be asked to reach as far as possible without stepping forward or touching the wall, while keeping their fist parallel to the tape measure. The point where the 3rd metacarpal reaches will be measured and recorded as the final reach distance.
Single-Leg Stance Test | In 2 weeks
  First, the participant will be asked which foot they prefer to stand on or which foot makes them feel more stable. Then, they will be instructed to distribute their weight evenly on both feet and, while maintaining this position, lift one foot off the ground. The timer will start as soon as the participant lifts their foot. The timer will be stopped if any signs of balance disturbance occur, such as the lifted foot making contact with the ground, the standing foot jumping, or the participant needing to support themselves in order to maintain balance.
Maximal exercise test | In 2 weeks
  Pre-exercise stress testing in asymptomatic adults with type 2 diabetes mellitus is a controversial topic. However, the American College of Sports Medicine recommends maximal exercise stress testing for individuals with diabetes over the age of 40, regardless of the presence of cardiovascular disease risk factors. In our study, the maximal exercise test will be performed on a treadmill under medical supervision to assess the risk of complications, and it will be conducted only before the exercise training program. The test will be carried out according to the Modified Bruce protocol.
Functional exercise capacity Functional Exercise Capacity | In 2 weeks
  Functional exercise capacity will be assessed using the 6-Minute Walk Test (6MWT). The participants will be instructed to walk at their maximum comfortable pace for 6 minutes along a 30-meter long, flat, and uninterrupted corridor. At the end of the test, the endpoint will be marked, and the total distance walked will be calculated.
Timed Up and Go Test (Cognitive) | In 2 weeks
  Participants will be asked to perform both the single-task and cognitive dual-task versions of the Timed Up and Go (TUG) test. In the single-task condition, participants will complete the TUG test without any secondary task. In the cognitive dual-task condition, participants will perform the TUG test while also engaging in a cognitive task, specifically subtracting 3 from 100 repeatedly during the walk.
Timed Up and Down Test (Standard-Cognitive) | In 2 weeks
  The Timed Up and Down Test (TUDT) is a measurement used to assess lower extremity functional muscle strength and balance. In the single-task condition, participants will perform the timed sit-to-stand test for 30 seconds without any secondary task. In the cognitive dual-task condition, participants will be asked to perform the sit-to-stand test while simultaneously subtracting 3 from 100 repeatedly.
Montreal Cognitive Assessment (MoCA) | In 2 weeks
  Cognitive function will be assessed using the Montreal Cognitive Assessment (MoCA). The MoCA is a reliable assessment tool that is particularly effective in testing cognitive levels in individuals with mild cognitive impairment and Alzheimer's disease. It is designed to evaluate various cognitive domains, including attention, memory, language, visuospatial abilities, executive functions, and orientation, providing a comprehensive measure of cognitive health. This tool is widely used in clinical settings for early detection and monitoring of cognitive decline.
Stroop Test | In 2 weeks
  The Stroop Test is a widely used psychological test to assess cognitive flexibility, selective attention, and the ability to inhibit cognitive interference. The test is based on the Stroop Effect, which refers to the delay in reaction time when the name of a color is written in a different color ink.
Diabetes-specific Quality of Life Scale (DQoL) | In 2 weeks
  The Diabetes-specific Quality of Life Scale (DQoL) is a self-report questionnaire designed to assess the quality of life (QoL) of individuals living with diabetes. It specifically focuses on how the disease and its management impact various aspects of daily life, such as emotional well-being, social functioning, and the physical burden of managing diabetes.
Processing Speed | In 2 weeks
  The processing speed will be evaluated by measuring the reaction time. To measure the reaction time, a FitLight Trainer (Fitlight Sports Corp., Canada) will be used. The FitLight Trainer is primarily used for training purposes and is also suitable for use with older individuals.
Muscle Strength | In 2 weeks
  The patients' overall muscle strength will be assessed using grip strength. The individuals' standard grip strengths will be measured with a Jamar hand dynamometer (Baseline Evaluation System, New York, USA). The measurement will be taken in the standardized test position as defined by the American Hand Therapy Association. Measurements will be taken on the dominant hand, with 3 repetitions and a 1-minute interval between each measurement, and the best value will be recorded in kg/force.
Pittsburgh Sleep Quality Index: PUKI | In 2 weeks
  The questionnaire is a widely used tool for assessing sleep quality. Developed in 1989 by Dr. Buysse and colleagues, this questionnaire evaluates individuals' sleep habits and sleep-related issues over the past month. The Pittsburgh Sleep Quality Index (PSQI) consists of 19 questions, covering factors such as sleep duration, time to fall asleep, sleep quality, insomnia, and daytime sleepiness. The score obtained from the questionnaire provides an overall assessment of a person's sleep quality.
Geriatric Depression Scale (GDS) | In 2 weeks
  In scoring the scale, 1 point is given for responses indicating depression, and 0 points are given for other responses. At the end of our study, individuals with a depression score above 14 will be considered depressed, while those with a score below 14 will be considered normal.
Activity-Specific Balance Confidence | In 2 weeks
  "Activity-specific balance confidence will be assessed using the Activity-Specific Balance Confidence (ABC) Scale (Powell & Myers, 1995). The ABC Scale, developed by Powell and Myers for the older population, assesses individuals' perceived level of confidence while performing daily living activities and the activities they feel can be safely performed without the risk of falling."
Biochemical Analysis | In 2 weeks
  Blood samples will be collected from patients with the supervision of a doctor to record their HbA1c and brain-derived neurotrophic factor (BDNF) levels before and after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: gizem mermerkaya, Principal Investigator — Bartın Unıversity
Locations (1):
- Bartın University, Bartın, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Villafaina S, Collado-Mateo D, Dominguez-Munoz FJ, Fuentes-Garcia JP, Gusi N. Impact of adding a cognitive task while performing physical fitness tests in women with fibromyalgia: A cross-sectional descriptive study. Medicine (Baltimore). 2018 Dec;97(51):e13791. doi: 10.1097/MD.0000000000013791. PMID 30572536
- [Background] Shellington EM, Reichert SM, Heath M, Gill DP, Shigematsu R, Petrella RJ. Results From a Feasibility Study of Square-Stepping Exercise in Older Adults With Type 2 Diabetes and Self-Reported Cognitive Complaints to Improve Global Cognitive Functioning. Can J Diabetes. 2018 Dec;42(6):603-612.e1. doi: 10.1016/j.jcjd.2018.02.003. Epub 2018 Mar 6. PMID 29884522
- [Background] Beauchet O, Dubost V, Aminian K, Gonthier R, Kressig RW. Dual-task-related gait changes in the elderly: does the type of cognitive task matter? J Mot Behav. 2005 Jul;37(4):259-64. PMID 15967751
- [Background] Tard C, Dujardin K, Girard A, Debaughrien M, Derambure P, Defebvre L, Delval A. How does visuospatial attention modulate motor preparation during gait initiation? Exp Brain Res. 2016 Jan;234(1):39-50. doi: 10.1007/s00221-015-4436-0. Epub 2015 Sep 10. PMID 26358126
- [Background] Park JH. Is Dual-Task Training Clinically Beneficial to Improve Balance and Executive Function in Community-Dwelling Older Adults with a History of Falls? Int J Environ Res Public Health. 2022 Aug 17;19(16):10198. doi: 10.3390/ijerph191610198. PMID 36011833
- [Background] Zhang J, Tam WWS, Hounsri K, Kusuyama J, Wu VX. Effectiveness of Combined Aerobic and Resistance Exercise on Cognition, Metabolic Health, Physical Function, and Health-related Quality of Life in Middle-aged and Older Adults With Type 2 Diabetes Mellitus: A Systematic Review and Meta-analysis. Arch Phys Med Rehabil. 2024 Aug;105(8):1585-1599. doi: 10.1016/j.apmr.2023.10.005. Epub 2023 Oct 22. PMID 37875170
- [Background] Callisaya ML, Daly RM, Sharman JE, Bruce D, Davis TME, Greenaway T, Nolan M, Beare R, Schultz MG, Phan T, Blizzard LC, Srikanth VK. Feasibility of a multi-modal exercise program on cognition in older adults with Type 2 diabetes - a pilot randomised controlled trial. BMC Geriatr. 2017 Oct 16;17(1):237. doi: 10.1186/s12877-017-0635-9. PMID 29037162